CLINICAL TRIAL: NCT01073202
Title: Effects of Ursodeoxycholic Acid on Graft Recovery Early After Adult Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFPH05B41
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Liver Transplantation; Ischemia-reperfusion Injury; Cholestasis
MeSH Terms: conditions — Reperfusion Injury; Cholestasis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- ursodeoxycholic acid (Active Comparator)
  Interventions: Drug: ursodeoxycholic acid
- identical-appearing placebo (Placebo Comparator)
  Interventions: Drug: identical-appearing placebo

INTERVENTIONS:
Drug: ursodeoxycholic acid — 13-15mg/kg/day, 250mg/capsule, given twice per day, within the first 4 weeks after liver transplantation
  Arms: ursodeoxycholic acid
Drug: identical-appearing placebo — 13-15mg/kg/day, 250mg/capsule, given twice per day, within the first 4 weeks after liver transplantation
  Arms: identical-appearing placebo

SUMMARY:
This study is designed to investigate the possible beneficial effects of UDCA on liver graft recovery early after adult liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All liver transplant patients in our center between May 2005 and April 2008 were potentially eligible for enrollment

Exclusion Criteria:

* Age less than 18 years
* Treatment with UDCA within one month before operation
* Inability to provide written informed consent prior to study entry
* Non-liver organ(s) failure prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Serum liver tests | within the first 4 weeks after liver transplantation
  Serum liver tests include serum levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transpeptidase (GGT), alkaline phosphatase (ALP) and total bilirubin (TB)

SECONDARY OUTCOMES:
Postoperative complications | within the first 4 weeks after liver transplantation
  Postoperative complications include rates of acute cellular rejection (ACR), drug-induced hepatotoxicity, vascular or biliary complications, recurrence of primary liver disease and death

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hai Peng, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Hertl M, Hertl MC, Kluth D, Broelsch CE. Hydrophilic bile salts protect bile duct epithelium during cold preservation: a scanning electron microscopy study. Liver Transpl. 2000 Mar;6(2):207-12. doi: 10.1002/lt.500060201. PMID 10719022
- [Background] Hertl M, Hertl MC, Kunkel P, Schilling S, Prevot B, Kluth D, Malago M, Broelsch CE. Tauroursodeoxycholate ameliorates reperfusion injury after pig liver transplantation. Transpl Int. 1999;12(6):454-62. doi: 10.1007/s001470050257. PMID 10654358
- [Background] Hertl M, Harvey PR, Swanson PE, West DD, Howard TK, Shenoy S, Strasberg SM. Evidence of preservation injury to bile ducts by bile salts in the pig and its prevention by infusions of hydrophilic bile salts. Hepatology. 1995 Apr;21(4):1130-7. PMID 7705788